CLINICAL TRIAL: NCT00002746
Title: A PHASE I TRIAL OF SUBCUTANEOUS, OUTPATIENT INTERLEUKIN-2 FOR PATIENTS WITH MYELODYSPLASTIC SYNDROME (MDS)
Brief Title: Interleukin-2 in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10469; UW-26-245-B; NCI-V96-0848
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety, tolerance, and maximum tolerated dose of subcutaneous interleukin-2 (aldesleukin; IL-2) in patients with myelodysplastic syndrome (MDS).
* Evaluate the hematologic effects of subcutaneous IL-2 in MDS.

OUTLINE: IL-2 will be administered in cycles of twice daily subcutaneous injections 7 days a week for 4 consecutive weeks. After each cycle the patient will be evaluated for response. The patient could continue IL-2 therapy for up to 12 cycles. There are 4 dose levels of IL-2. At each dose level 3 patients will be accrued sequentially.

Treatment with IL-2 should be continued until grade III toxicity or any side effects requiring hospitalization occurs. After the patient returns to baseline pretherapy values or grade I toxicity, the subject will resume IL-2 at 50% of the initial dose. If the patient again goes into grade III toxicity or is in need of hospitalization, IL-2 will be discontinued.

PROJECTED ACCRUAL: Between 12-24 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed myelodysplastic syndrome: Refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), refractory anemia with excess blasts (RAEB) or chronic myelomonocytic leukemia (CMML)
* No patients with refractory anemia with excess blasts in transformation (RAEB-t)

PATIENT CHARACTERISTICS:

Age:

* 15 and over

Performance status:

* Karnofsky 70-100

Hematopoietic:

* Platelet count greater than 20,000

Hepatic:

* Bilirubin less than 1.6 mg/dL
* SGOT less than 150 U/L

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No symptoms of coronary artery disease, congestive heart failure, edema, clinically manifest hypotension, presence of cardiac arrhythmias on EKG, or severe hypertension

Pulmonary:

* No significant pleural effusion, dyspnea at rest or severe exertional dyspnea

Other:

* No patients with nephrotic syndrome
* No uncontrolled infections or active peptic ulcer disease
* No serious intercurrent medical illness
* Not pregnant or nursing
* Adequate contraception required of all patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunosuppressive therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* At least 2 weeks since corticosteroid therapy
* At least 4 weeks since other endocrine therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1996-01; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Thompson, MD, Study Chair — Seattle Cancer Care Alliance
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States